CLINICAL TRIAL: NCT00283868
Title: A Prospective Study to Evaluate the Efficacy of a Remote Digital Observation Camera Protocol in the Evaluation and Thrombolytic Treatment of Acute Stroke Patients in the Remote Hospital Setting
Brief Title: Stroke Team Remote Evaluation Using a Digital Observation Camera
Acronym: STRokE DOC
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Brett C. Meyer, MD, UCSD Department of Neurology, UCSD Stroke Center
Other Study IDs: P50NS44148MEYER; P50NS044148 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2009-09

CONDITIONS: Stroke
Keywords: stroke; digital video; SPOTRIAS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Telemedicine: Patients randomized to this group were evaluated using the digital observation camera and DICOM evaluations for telemedicine
- Telephone: Patients randomized to this group were evaluated using telephone only and no use of the digital observation camera or DICOM

SUMMARY:
The purpose of this trial is to determine if an experimental remote video camera system is an effective way for a stroke specialist to evaluate stroke patients from a distant site.

DETAILED DESCRIPTION:
The Stroke Team Remote Evaluation Using a Digital Observation Camera (STRokE DOC) system is a digital video camera system that can transfer video and audio images from the clinic or emergency room to a distant (remote) place where a stroke specialist can review the images in real time (as they happen). This system uses site independent software to access the camera system from multiple locations. The study will determine if video consultation is superior to telephone consultation for remote evaluation or treatment of stroke patients, and the usefulness of this system in evaluating patients with suspected stroke symptoms. However, this method is being used in other fields of medicine for assistance in medical evaluations.

Participants will be randomly assigned to receive evaluation by either the video camera system or by telephone alone. For those assigned to the video camera system, the system will be activated and will record and transmit video and audio images to a stroke specialist located at a remote location. He/she may ask the participants questions relating to medical illnesses and current symptoms, and may also review laboratory tests and x-ray images using a computer, if available. The stroke specialist will also perform general physical and neurological examinations, which will take place by video camera with the assistance of a bedside physician who will perform the actual examinations.

For those participants assigned to the telephone-only consultation, the video system will not be activated, but the same procedure as above will be followed except the stroke specialist will not be able to see the participants or examine them using the video camera system. Participation in the study will last for the entire time the participants are in the hospital. Participants will be contacted by telephone by a study nurse 3 months post-stroke for a 10-minute interview regarding their current health. The total duration for individual participation is 3 months.

The study is part of the Specialized Program of Translational Research in Acute Stroke (SPOTRIAS), which allows researchers to enhance and initiate translational research that ultimately will benefit stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Symptoms consistent with acute stroke (ischemic or hemorrhagic)
* Acute presentation of stroke symptoms, per bedside physician discretion (onset generally less than 12 hours and likely less than 3 hours)

Exclusion Criteria:

* Unlikely to complete study through 90-day follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Stroke Patients
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2004-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Meyer, MD, Principal Investigator — UCSD Stroke Center
Locations (4):
- United States (4):
  - Pioneers Memorial Hospital, Brawley, California
  - El Centro Regional Medical Center, El Centro, California
  - University of California San Diego, San Diego, California
  - Twin Cities Community Hospital, San Luis Obispo, California

REFERENCES:
- [Background] Meyer BC, Lyden PD, Al-Khoury L, Cheng Y, Raman R, Fellman R, Beer J, Rao R, Zivin JA. Prospective reliability of the STRokE DOC wireless/site independent telemedicine system. Neurology. 2005 Mar 22;64(6):1058-60. doi: 10.1212/01.WNL.0000154601.26653.E7. PMID 15781827
- [Background] Crome O, Bahr M. Editorial comment--Remote evaluation of acute ischemic stroke: a reliable tool to extend tissue plasminogen activator use to community and rural stroke patients? Stroke. 2003 Oct;34(10):e191-2. doi: 10.1161/01.STR.0000095163.28915.B9. Epub 2003 Sep 18. No abstract available. PMID 14500919
- [Background] Patterson V. Teleneurology. J Telemed Telecare. 2005;11(2):55-9. doi: 10.1258/1357633053499840. PMID 15829048
- [Background] LaMonte MP, Bahouth MN, Hu P, Pathan MY, Yarbrough KL, Gunawardane R, Crarey P, Page W. Telemedicine for acute stroke: triumphs and pitfalls. Stroke. 2003 Mar;34(3):725-8. doi: 10.1161/01.STR.0000056945.36583.37. Epub 2003 Jan 30. PMID 12624298
- [Background] Schwamm LH, Rosenthal ES, Hirshberg A, Schaefer PW, Little EA, Kvedar JC, Petkovska I, Koroshetz WJ, Levine SR. Virtual TeleStroke support for the emergency department evaluation of acute stroke. Acad Emerg Med. 2004 Nov;11(11):1193-7. doi: 10.1197/j.aem.2004.08.014. PMID 15528584
- [Background] Audebert HJ, Kukla C, Clarmann von Claranau S, Kuhn J, Vatankhah B, Schenkel J, Ickenstein GW, Haberl RL, Horn M; TEMPiS Group. Telemedicine for safe and extended use of thrombolysis in stroke: the Telemedic Pilot Project for Integrative Stroke Care (TEMPiS) in Bavaria. Stroke. 2005 Feb;36(2):287-91. doi: 10.1161/01.STR.0000153015.57892.66. Epub 2004 Dec 29. PMID 15625294
- [Background] Wiborg A, Widder B; Telemedicine in Stroke in Swabia Project. Teleneurology to improve stroke care in rural areas: The Telemedicine in Stroke in Swabia (TESS) Project. Stroke. 2003 Dec;34(12):2951-6. doi: 10.1161/01.STR.0000099125.30731.97. Epub 2003 Nov 20. PMID 14631092
- [Background] Wang S, Gross H, Lee SB, Pardue C, Waller J, Nichols FT 3rd, Adams RJ, Hess DC. Remote evaluation of acute ischemic stroke in rural community hospitals in Georgia. Stroke. 2004 Jul;35(7):1763-8. doi: 10.1161/01.STR.0000131858.63829.6e. Epub 2004 May 27. PMID 15166386
- [Derived] Demaerschalk BM, Raman R, Ernstrom K, Meyer BC. Efficacy of telemedicine for stroke: pooled analysis of the Stroke Team Remote Evaluation Using a Digital Observation Camera (STRokE DOC) and STRokE DOC Arizona telestroke trials. Telemed J E Health. 2012 Apr;18(3):230-7. doi: 10.1089/tmj.2011.0116. Epub 2012 Mar 8. PMID 22400970
- [Derived] Meyer BC, Raman R, Hemmen T, Obler R, Zivin JA, Rao R, Thomas RG, Lyden PD. Efficacy of site-independent telemedicine in the STRokE DOC trial: a randomised, blinded, prospective study. Lancet Neurol. 2008 Sep;7(9):787-95. doi: 10.1016/S1474-4422(08)70171-6. PMID 18676180
- [Derived] Meyer BC, Raman R, Chacon MR, Jensen M, Werner JD. Reliability of site-independent telemedicine when assessed by telemedicine-naive stroke practitioners. J Stroke Cerebrovasc Dis. 2008 Jul-Aug;17(4):181-6. doi: 10.1016/j.jstrokecerebrovasdis.2008.01.008. PMID 18589337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment completed in 4/07
Pre-assignment Details: There were 11 initial "run-in" patients used to validate the system but these patients were excluded from the final analysis. There was also 1 patient removed from analysis because of a protocol violation (age < 18) so this patient was excluded rom any analysis (Initial patients=234. 11 Run in=223. 1 removed=222. This accounts for final numbers)
Groups:
- Telephone: Patients randomized to this group were only evaluated using telephone and were not evaluated using the digital observation camera or DICOM
Period: Overall Study
Arm/Group | Telemedicine | Telephone
Started | 111 | 111
Completed | 104 | 103
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemedicine | Telephone | Total
Number analyzed (Participants) | 111 | 111 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 38 | 36 | 74.0
  >=65 years | 73 | 75 | 148.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (14.5) | 69 (14.9) | 69.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114.0
  Male | 54 | 54 | 108.0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 111 | 222.0

OUTCOME MEASURES:

1. Primary Outcome: Appropriateness of Decision to Treat or Not Treat With Thrombolytics
Description: This primary measure assesses the appropriateness of decision to treat or not treat with thrombolytics for patients presenting potentially within 3 hours of symptom onset.
  Appropriateness was assessed using a centralized adjudicating committee, 3 levels of data availability, and an independent medical monitor assessment. The case was presented to the adjudicating committee (blinded to randomization arm) and the committee reviewed patient records (also blinded to randomization arm) to assess whether decision was "appropriate" to give or not give rt-PA.
Time Frame: potentially within 3 hours of symptom onset
Population: Of the original 234 patients, 11 were run in patients and were not randomized and 1 was removed from any analysis due to a protocol violation resulting in the total 222 patients analyzed. There were 7 lost to follow up in telemedicine and 8 lost to follow up in telephone resulting in 104 analyzed in telemedicine and 103 analyzed in telephone.
Measure: Number; unit: percentage of participants
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 104 | 103
percentage of participants | 98 | 82

2. Secondary Outcome: Percentage of Participants With Intracerebral Hemorrhage (ICH)
Description: Intracerebral Hemorrhage (ICH) rate at 36 hours. This was assessed by determining whether there was an intracerebral hemmorhage via telephone contact to the hospital where the patient was located. Any follow up imaging (head CT or MRI) was reported to the investigator team for presence of hemorrhage.
Time Frame: 36 hours
Measure: Number; unit: Percentage of participants
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 104 | 103
Percentage of participants | 7 | 8

3. Secondary Outcome: Percentage of Total Thrombolytic Administrations
Description: This measure assesses the number of total thrombolytic administrations that were given. This was to measure whether there were more participants treated with thrombolytics in one arm of the trial or the other.
Time Frame: potentially within 3 hours of symptom onset
Measure: Number; unit: Percentage of participants
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 104 | 103
Percentage of participants | 28 | 23

4. Secondary Outcome: Time to Treatment Decision for Administration of Thrombolytics
Description: time to decision (consult onset to decision). This measure was meant to assess how long it took to do the evaluation.
Time Frame: potentially within 3 hours of symptom onset
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 104 | 103
Minutes | 32 (17) | 23 (24)

5. Secondary Outcome: Percentage of Evaluations With Technical Observations
Description: Technical Observations: This measure was designed to assess the percentage of evaluations where there were technical observations (difficulties with using the technology) noted by the consultant who performed the evaluation (either telemedicine evaluation or telephone evaluation) in each arm of the trial.
Time Frame: Time of consultation
Measure: Number; unit: Percentage of Evaluations
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 104 | 103
Percentage of Evaluations | 0 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No